CLINICAL TRIAL: NCT05506202
Title: Individual Basic Body Awareness Therapy (BBAT) as an add-on Treatment for Dyspnea Self-management in Patients With Chronic Obstructive Pulmonary Disease (COPD) - a Quantitative and Qualitative Study
Brief Title: Basic Body Awareness Therapy (BBAT) for Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North District Hospital (Other)
Responsible Party: Principal Investigator, Mo Kim Chung, Physiotherapist I, North District Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022.316
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Basic body awareness therapy; Chronic obstructive pulmonary disease; Dyspnea; Self-management; Physiotherapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): In intervention group, one extra physiotherapeutic intervention, Basic Body Awareness Therapy (BBAT), will be provided before ending each visit (on top of basic and advanced respiratory physiotherapy interventions as control group). Each BBAT last for 30-45 minutes. Therapist will verbally guide patients to perform twelve simple and soft movements, including lying, sitting, standing, walking and relational movements in a quiet and secured environment. Therapist will allow patients to explore the movement and the experience. Therapist will also guide patients in shifting focus between balance, free breathing and mental awareness Following principles in BBAT, BBAT movements will be selected for patients as home exercises.
  Interventions: Other: Individual basic body awareness therapy; Other: Respiratory physiotherapy interventions
- Control group (Active Comparator): Both basic and advanced respiratory physiotherapy interventions, including respiratory muscles training, breathing techniques, bronchial hygiene maintenance, assisting in non-invasive ventilation therapy and oxygen therapy titration, are provided according to assessment findings. There is an eight-week training program for both groups, therapist will provide one home visit per week and continuously for eight weeks for each patient.
  Interventions: Other: Respiratory physiotherapy interventions

INTERVENTIONS:
Other: Individual basic body awareness therapy — Basic Body Awareness Therapy (BBAT) is a physiotherapeutic intervention directed toward patients' functional movement quality. The development of BBAT was based on the hypothesis of persons' lacking contact with and lacking awareness on their own body, with their inner life, external environment and in the relation to other persons. Thus, it leads to dysfunctional movement, pain and other body functions. BBAT focus on multi-perspective within a person including physical, physiological, psycho-social-cultural and existential perspectives. It directs patients to be "aware", guides patients to have mental contact with their body, monitors internal sensations and external environment, and thus, to enhance the self-regulated behavior and positive emotional state.
  Arms: Intervention group
Other: Respiratory physiotherapy interventions — Comprehensive physical and psycho-social assessment and treatments are included. Both basic and advanced respiratory physiotherapy interventions, including respiratory muscles training, breathing techniques, bronchial hygiene maintenance, assisting in non-invasive ventilation therapy and oxygen therapy titration, are provided according to assessment findings.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a burden to health care and economic systems globally, to manage this preventable and treatable disease, different pharmacological and non-pharmacological interventions were shown to be effective.

Chronic and progressive dyspnea, cough and sputum production are the characteristic symptoms of COPD. The most commonly encountered symptom in patients with COPD is dyspnea, it is a subjective experience of breathing discomfort . It causes impact on patient's health status, sleep quality, anxiety and depression level. Therefore, skills transfer in self-managing major symptoms are crucial to prevent negative consequences, and as suggested by Global Initiative for Chronic Obstructive Lung Disease (GOLD), managing symptoms and to prevent future risk of exacerbations is important for stable COPD cases.

Basic Body Awareness Therapy (BBAT) is a physio-therapeutic intervention directed toward patients' functional movement quality. The development of BBAT was based on the hypothesis of persons' lacking contact with and lacking awareness on their own body, with their inner life, external environment and in the relation to other persons. Thus, it leads to dysfunctional movement, pain and other body functions. BBAT focus on multi-perspective within a person including physical, physiological, psycho-social-cultural and existential perspectives. It directs patients to be "aware", guides patients to have mental contact with their body, monitors internal sensations and external environment, and thus, to enhance the self-regulated behavior and positive emotional state.

There are three key components in practicing BBAT, namely balance, free breathing and mental awareness. Evidence shown that the effect of BBAT is significant in improving physical and psycho-social well-being in patients with different physical and mental disorders. Now, there is absence of evidence in applying BBAT in managing cases with respiratory diseases, especially for those with prominent symptoms of dyspnea (for example COPD cases).

The objectives of this study are (1) to evaluate individual BBAT as an add-on treatment in patients with COPD, (2) to understand COPD patients' experience through participating in individual Basic Body Awareness Therapy (BBAT).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with COPD (ICD-9-CM 496.X) AND
* Ability to stand independently without aids, AND
* Subjectively experienced dyspnea, AND
* Ability to listen, speak, read and understand Chinese.

Exclusion Criteria:

* Patients with acute exacerbation of COPD within one-month, OR
* Patients with medical disorders possibly causing dyspnea (for example asthma, heart failure, etc.), OR
* Patients with major psychiatric or cognitive disorders, OR
* Patients refusal

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Modified Medical Research Council scale for breathlessness | 2 months
  mMRC is used to establish patients' baseline functional impairment due to dyspnea, scale from 0 to 4, with 0 indicates only get breathless with strenuous exercise, and 4 indicates too breathless to leave the house or I am breathless when dressing/undressing
Dyspnoea-12 (Chinese version) | 2 months
  Dyspnoea-12 is used to measure patients' dyspnea severity, scale range, 0-36, with a high score indicating worse dyspnea
St. George's Respiratory Questionnaire (Chinese version) | 2 months
  St. George's Respiratory Questionnaire is used to measure patients' health-related quality of life, Scores range from 0 to 100, with higher scores indicating more limitations.
COPD Self-Efficacy Scale (Chinese version) | 2 months
  COPD Self-Efficacy Scale contains 34 items, each item rated by Likert 5-level score ranges from 1 point (completely unconfident) to 5 points (completely confident).
6 minutes walking test | 2 months
  6 minutes walking test is used to assess patients' functional capacity, the outcome is measuring distance covered and counts in meters, with higher meters covered indicates a better functional capacity

CONTACTS AND LOCATIONS:
Locations (1):
- North District Hospital, Hong Kong, Hong Kong